CLINICAL TRIAL: NCT07293026
Title: Clinical Study on the Efficacy of Abdominal Acupuncture in Promoting Gastrointestinal Function Recovery After Gynecological Laparoscopic Surgery
Brief Title: Abdominal Acupuncture for Gastrointestinal Function Recovery After Gynecologic Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mengyao Han (Other)
Responsible Party: Sponsor-Investigator, Mengyao Han, Researcher, Guangdong Provincial Hospital of Traditional Chinese Medicine
Organization: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YF2023-435
Record Dates: First submitted 2025-10-02; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Complications; Postoperative Gastrointestinal Dysfunction (POGD); Postoperative Ileus
Keywords: abdominal acupuncture; gastrointestinal function; quality of life; Postoperative Gastrointestinal Dysfunction; Postoperative Ileus; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal acupuncture treatment group (Experimental): In addition to standard postoperative care, patients received abdominal acupuncture. In the supine position, acupoints were localized proportionally from the umbilicus (CV8): 8 cun upward to CV16, 5 cun downward to the pubic symphysis, and 6 cun laterally. After aseptic skin preparation, disposable sterile needles were inserted perpendicularly. Primary points were needled at the Di level (1.0-1.5 cun) for visceral regulation and secondary points at the Ren level (0.5-1.0 cun) for peripheral stimulation. Gentle rotation was applied without lifting or thrusting, and deqi was not required. Needles were retained for 30 minutes with concurrent infrared warming. After withdrawal, sterile compression prevented bleeding. The first session was administered 4-6 hours postoperatively, followed by one daily on postoperative days 1-4, totaling five sessions. Clinical status was documented throughout.
  Interventions: Procedure: Abdominal acupuncture; Other: Standard postoperative management protocol
- control group (Active Comparator): The standardized postoperative management protocol consists of the following components:
  1. Early oral intake: patients may commence a liquid diet 6 hours after surgery, advance to a semi-liquid diet following the passage of flatus, and transition to a regular diet after bowel movement.
  2. Early mobilization: patients are encouraged to turn in bed and initiate physical activity as early as 6 hours postoperatively, and to ambulate as soon as their condition permits.
  3. Adequate fluid supplementation.
  4. Maintenance of fluid-electrolyte and acid-base balance.
  5. Prophylactic antibiotic therapy to prevent infection.
  6. Early removal of urinary catheters, drainage tubes, and other indwelling devices.
  7. Postoperative analgesia: implementation of a multimodal pain management strategy.
  8. In critically ill patients, supplemental oxygen and continuous electrocardiographic monitoring are required.
  Interventions: Other: Standard postoperative management protocol

INTERVENTIONS:
Procedure: Abdominal acupuncture — Patients were positioned supine with the abdomen exposed. Acupoint selection and localization followed Abdominal Acupuncture Therapy standards, with proportional measurements taken from the umbilicus (CV8): 8 cun upward to CV16, 5 cun downward to the pubic symphysis, and 6 cun laterally. After hand hygiene and aseptic skin preparation, disposable sterile needles were inserted perpendicularly. Primary acupoints were needled at the Di level (1.0-1.5 cun) targeting visceral disorders, and secondary acupoints at the Ren level (0.5-1.0 cun) for peripheral regulation. Gentle rotation was employed without lifting/thrusting, and deqi induction was not required. Needles were retained for 30 minutes with concurrent infrared warming therapy. Post-treatment, needles were withdrawn with sterile compression applied to prevent bleeding. The first session was given 4-6 hours postoperatively, followed by one session daily on postoperative days 1-4, for a total of five sessions.
  Other Names: acupuncture; Abdominal acupuncture treatment; Bo's Abdominal Acupuncture
  Arms: Abdominal acupuncture treatment group
Other: Standard postoperative management protocol — Multimodal perioperative care including early oral intake, early mobilization, fluid and electrolyte balance, prophylactic antibiotics, device removal, multimodal analgesia, and supportive monitoring; gastrointestinal prokinetics, enemas, and herbal medicines prohibited.

SUMMARY:
Current research on the role of abdominal acupuncture in promoting postoperative gastrointestinal recovery remains limited, characterized by a lack of large-scale, standardized clinical trials, particularly with respect to long-term outcomes. This study, grounded in a rigorous randomized controlled trial design, investigates the clinical efficacy of abdominal acupuncture in enhancing gastrointestinal function following gynecologic laparoscopic surgery. The findings aim to provide a scientific foundation for improving postoperative quality of life, optimizing recovery pathways in gynecology, and identifying safer, simpler, and more effective therapeutic options. In addition, this work offers theoretical support and practical evidence to advance the clinical integration and broader application of traditional Chinese therapeutic approaches in modern surgical rehabilitation, underscoring its significant clinical value.

DETAILED DESCRIPTION:
This single-center, randomized, parallel-group clinical trial evaluates the adjunctive use of Bo's abdominal acupuncture in women undergoing laparoscopic total hysterectomy at Guangdong Provincial Hospital of Chinese Medicine. The trial is designed to test whether adding abdominal acupuncture to standardized postoperative care can enhance gastrointestinal recovery and is safe in this setting. The protocol was approved by the institutional ethics committee. Eligible participants are randomized 1:1 using an independently generated, concealed allocation sequence (sequentially numbered, opaque, sealed envelopes). Because of the nature of the intervention, treating acupuncturists are not blinded, while outcome assessors and data analysts remain blinded to group assignment.

All participants receive standardized postoperative care per institutional pathways, and therapies that directly affect gastrointestinal motility are restricted unless prespecified rescue criteria are met. Participants assigned to the intervention arm receive Bo's abdominal acupuncture beginning 4-6 hours after surgery and once daily on postoperative days 1-4 (five sessions in total). Treatment follows a standardized technique grounded in pattern differentiation, delivered with sterile single-use needles and approximately 30 minutes of needle retention; full procedural details are provided in the Interventions section of this record. Outcomes, instruments, and time frames are prespecified in the Outcome Measures module; the primary endpoint is time to first passage of flatus, and secondary measures encompass gastrointestinal recovery, adverse events and postoperative complications, inflammatory biomarkers, pain, and gastrointestinal quality of life. Safety is monitored throughout with reporting per institutional policy. Statistical analyses will follow an intention-to-treat approach where feasible, using appropriate parametric or nonparametric tests for continuous variables, chi-square or Fisher exact tests for categorical variables, and repeated-measures models for longitudinal data, with two-sided α=0.05 and effect estimates reported with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients who underwent gynecologic laparoscopic total hysterectomy under general anesthesia;
2. Age between 18 and 65 years;
3. Surgical duration ranging from 0.5 to 4.5 hours;
4. Anesthesia duration ranging from 1 to 5 hours;
5. Willingness to receive acupuncture therapy without a history of adverse reactions such as needle syncope;
6. Provision of signed informed consent.

Exclusion Criteria:

1. Patients with comorbid conditions that may affect gastrointestinal function, including intestinal obstruction or space-occupying lesions of the digestive system;
2. Patients with severe systemic diseases, including hepatic or renal failure, cardiovascular or cerebrovascular disorders, infectious diseases such as HIV/AIDS, or severe psychiatric illness;
3. Individuals with a history of adverse reactions to acupuncture, including needle syncope;
4. Patients with local skin damage, rashes, or ulcers at the proposed acupoint sites;
5. Patients concurrently enrolled in other clinical studies.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Time to first postoperative passage of flatus | From the end of surgery until the first documented passage of flatus; assessed through postoperative Day 5 or hospital discharge, whichever occurs first.
  Elapsed time from the end of laparoscopic gynecologic surgery to the first documented passage of flatus; patient-reported and nurse-confirmed. Time is recorded in hours and minutes. Per protocol, rescue therapy may be used if no flatus by postoperative Day 3.

SECONDARY OUTCOMES:
Time to first postoperative bowel movement | From the end of surgery until the first documented bowel movement; assessed through postoperative Day 5 or hospital discharge, whichever occurs first.
  Elapsed time from the end of laparoscopic gynecologic surgery to the first documented bowel movement; patient-reported and nurse-confirmed. Time is recorded in hours and minutes. Rescue therapy may be used if no bowel movement by postoperative Day 3.
restoration of bowel sounds | From the end of surgery until the first detection of normal bowel sounds; assessed every 8 hours through postoperative Day 5 or hospital discharge, whichever occurs first.
  Elapsed time from the end of surgery to the first auscultated normal bowel sounds (defined as 4 or more sounds per minute in all four quadrants). Auscultation is performed every 8 hours until recovery.
Incidence of postoperative gastrointestinal dysfunction | From the day of surgery through postoperative Day 5 or hospital discharge, whichever occurs first.
  Proportion of participants with gastrointestinal dysfunction-related complications (abdominal bloating/pain, nausea, vomiting, diarrhea, or postoperative ileus). Events are confirmed by a physician or nursing staff.
Inflammatory markers | Each parameter was assessed once preoperatively, on the day of surgery prior to treatment, and on postoperative Day 5.
  Inflammatory markers included C-reactive protein (CRP), serum interleukin-6 (IL-6), serum tumor necrosis factor-α (TNF-α), and the systemic immune-inflammation index [SII, SII = (platelet count × neutrophil count) / lymphocyte count].
  Each parameter was assessed once preoperatively, on the day of surgery prior to treatment, and on postoperative Day 5.
Pain assessment | Day 0 (day of surgery) and Postoperative Days 1 through 5; or until hospital discharge if earlier.
  Abdominal pain intensity will be assessed using the Visual Analog Scale for Pain (VAS), a 10-centimeter horizontal line anchored at 0 = no pain and 10 = worst imaginable pain. Scores range from 0 to 10; higher scores indicate worse pain. Assessments will be performed twice on the day of surgery (before and after the first acupuncture session) and once daily on Postoperative Days 1 through 5.
Gastrointestinal Symptom Score | Day 0 (day of surgery; pre-intervention assessment) and Postoperative Days 1 through 5; assessed once daily or until hospital discharge if earlier.
  Adapted from the Perioperative Clinical Evaluation Standards for Gastrointestinal Motility (Guangdong Provincial Standard). Composite of nine items: flatus (present=15; absent=0), defecation (present=15; absent=0), abdominal distension/pain (none=10; mild=5; intolerable=0), bowel sounds (normal=10; reduced=5; absent=0), nausea (none=10; mild with activity only=5; intermittent or persistent at rest=0), vomiting (none=10; 1-2/day=5; ≥3/day=0), diarrhea (none=10; 1-2/day=5; ≥3/day=0), surgical incision (well-approximated without redness/swelling/pain=10; any of these, fat liquefaction, or dehiscence=0), and body temperature (≤37.5°C=10; 37.5-<39.0°C=5; ≥39.0°C=0). Total score 0-100; higher scores indicate better gastrointestinal function. Normal bowel sounds are defined as ≥4 sounds/min in all quadrants. Episode counts refer to the prior 24 hours for vomiting/diarrhea. Assessments are performed by trained staff and recorded in case report forms.
Gastrointestinal quality of life assessment | Day 0 (day of surgery; pre-intervention baseline), Postoperative Day 5 (or at hospital discharge if earlier), and approximately Postoperative Day 19 (14 days after the final treatment; allowable window ±2 days).
  Health-related quality of life will be measured using the Gastrointestinal Quality of Life Index (GIQLI). The GIQLI is a 36-item questionnaire covering gastrointestinal symptoms, physical function, emotional status, social function, and the effect of treatment. Each item is scored 0-4, yielding a total score of 0-144 points; higher scores indicate better health-related quality of life. The recall period is the past week (one-week recall); the items and scoring follow the original instrument.

OTHER OUTCOMES:
Adverse Events | From the day of surgery (Day 0) through Postoperative Day 19 (14 days after the final treatment session), including the treatment period and follow-up.
  All adverse events were monitored from surgery to postoperative Day 19, including needle-related events (needle stagnation, syncope, breakage, hematoma, infection) and any other AEs. Each was promptly managed and recorded in CRFs.

CONTACTS AND LOCATIONS:
Overall Officials: YI Chen, Ph.D, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Can be shared after research paper is published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It is not yet determined. The relevant content can be shared after the paper is published.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT07293026/Prot_000.pdf
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT07293026/ICF_001.pdf